CLINICAL TRIAL: NCT03364179
Title: IssuEs in Palliative Care for People in Advanced and Terminal Stages of Young-onset and Late-Onset Dementia in GErmany (EPYLOGE-Study)
Brief Title: IssuEs in Palliative Care for People in Advanced and Terminal Stages of Young-onset and Late-Onset Dementia in GErmany
Acronym: EPYLOGE
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Deutsche Alzheimer Gesellschaft (Unknown); Centre Hospitalier Universitaire Vaudois (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Janine Diehl-Schmid, Clinical Professor, Principle Investigator, Technical University of Munich
Other Study IDs: PALLVFKS022EPYLOGE
Record Dates: First submitted 2017-10-16; First posted 2017-12-06 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Advanced Dementia Stages; Palliative Care
Keywords: dementia; young onset dementia; quality of death; late onset dementia; palliative care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- young onset dementia
- late onset dementia

SUMMARY:
From a scientific view, palliative care issues in dementia are neglected in Germany. Neither in Germany nor internationally research has been conducted on palliative care issues in young onset dementia (YOD), although significant differences compared to late onset dementia (LOD) are expected. Most international studies have focused on patients in long term care (LTC) facilities but have neglected patients that are cared for at home. We hypothesize that in advanced and terminal stages of YOD and LOD unmet care needs exist and that they differ between YOD and LOD. By prospectively assessing and surveying 200 patients with YOD and LOD in advanced stages who are cared for in LTC facilities and at home and investigating circumstances of death of 100 YOD- and LOD-patients, it is possible 1) to describe symptoms and management, health care utilization, palliative care provision, quality of life and death, elements of advance care planning, family caregivers' needs and satisfaction; 2) to compare YOD and LOD; 3) to develop expert-consensus recommendations derived from study results for the improvement and implementation of strategies and interventions for palliative care provision. 4) to communicate the recommendations nationally and internationally in order to improve and adapt guidelines, to implement the recommendations into daily practice and to give a basis and perspectives for future research projects; to communicate the results to patients and their families in order to counsel and support them in their decision making processes and their dialogue with professional caregivers and physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patient with moderate or severe dementia (CDR = 2 or 3)
* Patient lives at home or in long term care
* Patient has got a family caregiver > 18 years
* Family caregiver has sufficient knowledge of German language
* Written informed consent of family caregiver
* Written informed consent of patient or legal representative, respectively
* Documents of legal representative/ Power of attorney

Exclusion criteria

• at least one inclusion criterion is not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from young onset and late onset dementia in advanced and terminal stages who live in LTC facilities or at home and their family caregivers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-08-19 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
patient´s quality of life in late stage dementia | Baseline
  Quality of ife in late-stage dementia scale (QUALID-Scale): 11 questions, Score 1 to 5 each, total sum score range 11 to 55, 11 means highest quality of life
patient´s comfort of dying with dementia | Assessment B at the latest 4 months after patient's death
  Comfort assessment of dying with dementia (CAD-EOLD)-Scale: Subscale of End of Life in Dementia Scale (EOLD), 14 symptoms/ conditions during patient´s dying process to be rated by proxy, Score 1-3 each. Total sum score range 14 to 42. 42 means highest level of comfort during dying process.

SECONDARY OUTCOMES:
symptoms and symptom management in late-stage dementia and during the dying process | Assessment A (study inclusion, patient is alive) and Assessment B (as soon as possible after patient´s death, at the latest 4 months after death)
  adapted version of End of Life in Dementia -Symptom Management scale (SM-EOLD); patient´s examination; assessment of drug treatment and non-medical therapies by evaluation of medical files
palliative care provision in late-stage dementia and during the dying process | Assessment A (inclusion, patient is alive) and Assessment B (as soon as possible after patient´s death, at the latest 4 months after death)
  semi-structured interviews with the caregiver to assess the status quo of (palliative) care issues (e.g. availability of general outpatient palliative care (AAPV), specialized outpatient palliative care (SAPV) or palliative care nurses; description of LTC setting; caregivers´experiences with palliative care)
health care utilization in late-stage dementia and during the dying process | Assessment A (inclusion, patient is alive) and Assessment B (as soon as possible after patient´s death, at the latest 4 months after death)
  semi-structured interviews with the caregivers
Caregivers' problems, challenges, barriers, needs, preferences in late-stage dementia and during the dying process | Assessment A (inclusion, patient is alive) and Assessment B (as soon as possible after patient´s death, at the latest 4 months after death)
  open questions to the family caregiver
family caregivers' burden and coping | Assessment A (inclusion, patient is alive) and Assessment B (as soon as possible after patient´s death, at the latest 4 months after death)
  various scales, e.g. the adapted version of Caregiver Strain Index (CSI)
family caregivers´satisfaction with care | Assessment A (inclusion, patient is alive) and Assessment B (as soon as possible after patient´s death, at the latest 4 months after death)
  various scales, e.g. the adapted version of End of life in dementia-Satisfaction with Care, (SWC-EOLD)

CONTACTS AND LOCATIONS:
Locations (1):
- Zentrum für kognitive Störungen, Psychiatrische Klinik und Poliklinik, Klinikum Rechts der Isar, TU München, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Diehl-Schmid J, Hartmann J, Rossmeier C, Riedl L, Forstl H, Egert-Schwender S, Kehl V, Schneider-Schelte H, Jox RJ. IssuEs in Palliative care for people in advanced and terminal stages of Young-onset and Late-Onset dementia in GErmany (EPYLOGE): the study protocol. BMC Psychiatry. 2018 Aug 31;18(1):271. doi: 10.1186/s12888-018-1846-0. PMID 30170575
- [Derived] Diehl-Schmid J, Rossmeier C, Slawik T, Hartmann J, Riedl L, Kehl V. Home Care of People With Advanced Late-Onset and Young-Onset Dementia Living in Germany. Alzheimer Dis Assoc Disord. 2025 Oct-Dec 01;39(4):263-268. doi: 10.1097/WAD.0000000000000687. Epub 2025 Nov 14. PMID 41233710
- [Derived] Riedl L, Kiesel E, Hartmann J, Fischer J, Rossmeier C, Haller B, Kehl V, Priller J, Trojan M, Diehl-Schmid J. A bitter pill to swallow - Polypharmacy and psychotropic treatment in people with advanced dementia. BMC Geriatr. 2022 Mar 16;22(1):214. doi: 10.1186/s12877-022-02914-x. PMID 35296254
- See also: EPYLOGE. Eine Studie zur Palliativversorgung bei Demenz in Deutschland — https://www.zks.psykl.mri.tum.de/aktuelles/aktuelle-meldung/news/epyloge/?tx_news_pi1%5Bcontroller%5D=News&tx_news_pi1%5Baction%5D=detail&cHash=9416566d7fb15872ce704b354d1d3f18